CLINICAL TRIAL: NCT02513134
Title: Intraocular Lens Power Calculation Using Pre- and Intra-operative
Brief Title: Intraocular Lens Power Calculation Using Pre- and Intra-operative Measurements
Status: Completed | Type: Observational
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr. MBA, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Other Study IDs: OC3; OC3 (Registry Identifier: OC3)
Record Dates: First submitted 2014-06-02; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Cataract
Keywords: IOL power calculations; Intraoperative; OCT; Refractive outcome; Biometry
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recently a prototype of a combination of an anterior segment OCT (VISANTE; Carl Zeiss Meditec AG) and an operating microscope (OPMI 200; Carl Zeiss Meditec AG) was introduced that allows measurements of the crystalline lens as well as the lens capsule itself after removing the crystalline lens of cataract patients intra-operatively. This device uses OCT technology to create high resolution B-scans (=images) of the anterior segment of the eye. The OCT was shown to be highly reproducible for ACD measurements pre-operatively 12 and small changes of the IOL/crystalline lens can be detected 13.

In a previous study (EK-10-125-0710) that was recently published in the journal "Investigative Ophthalmology & Visual Science" it was shown that intra-operative measurements of the anterior lens capsule improve the refractive outcome theoretically.14 However, in this previous study conventional eye models were used for IOL power calculation and only the intra-operative measurement replaced pre-operative ACD measurements.

Aim of this study is to observe, whether the postoperative refractive outcome could be improved theoretically by using both pre- and intra-operative measurements for retrospective IOL power calculation with new eye models.

DETAILED DESCRIPTION:
Since the introduction of optical biometry 1 (IOLMaster, Carl Zeiss Meditec AG, Jena, Germany), as a reliable non-contact measurement of the axial eye length the influence of the error of axial length measurement on the refractive error decreased from over 50% (when measured with applanation ultrasound) to 36%. The mean error of corneal power measurement is approximately 22% 2. These results show that the estimation of the post-operative intra-ocular lens (IOL) position and therefore the estimated anterior chamber depth (ACD) is nowadays the main source of error (35% 3 to 42% 2) in IOL power calculation and therefore for the refractive outcome of the patients after cataract surgery. Early IOL power calculation formulae, such as the Binkhorst I formula 4, used a fixed ACD value to predict the position of the IOL, but the refractive results were not appropriate, because the post-operative position of the IOL varied significantly between patients. Later observations showed a correlation between the axial eye length and the post-operative ACD (longer=more myopic eyes showed a larger ACD post-operatively). 5 These correlations were taken into account in later developed formulas (such as the Binkhorst II formula). Olsen et al. 6 measured the post-operative ACD and substituted the predicted post-operative ACD with the true, post-operative ACD in each case. The result after correcting the IOL position was a highly accurate IOL power calculation, where no fudge factors were needed. Nowadays the pre-operatively measured ACD is taken into account for several IOL power calculation formulas, such as the Haigis formula, the Holladay II formula and the Olsen formula. However, this new generation of formulas use the pre-operative ACD, without considering the thickness of the crystalline lens. The ACD is measured as the distance between the anterior surface of the cornea (anatomically correct would be the posterior surface of the cornea, but in an optical context, as in IOL power calculations, the anterior surface is used) and the anterior surface of the crystalline lens 2. Therefore the thickness of the crystalline lens has a significant impact on the predicted post-operative position of the IOL. This parameter was first taken into account by Olsen 7 and later modified by Norrby 8, 9. It should be mentioned that IOL power calculations developed from theoretical calculations based on Gaussian optics 10 to regression formulas, such as the SRK formula 11 that uses retrospective data of a large number of patients. All these findings suggest that proper measurements not only of the dimensions of the crystalline lens but also of the lens capsule after removing the crystalline lens are necessary to improve IOL power calculation.

Recently a prototype of a combination of an anterior segment OCT (VISANTE; Carl Zeiss Meditec AG) and an operating microscope (OPMI 200; Carl Zeiss Meditec AG) was introduced that allows measurements of the crystalline lens as well as the lens capsule itself after removing the crystalline lens of cataract patients intra-operatively. This device uses OCT technology to create high resolution B-scans (=images) of the anterior segment of the eye. The OCT was shown to be highly reproducible for ACD measurements pre-operatively 12 and small changes of the IOL/crystalline lens can be detected 13.

In a previous study (EK-10-125-0710) that was recently published in the journal "Investigative Ophthalmology & Visual Science" it was shown that intra-operative measurements of the anterior lens capsule improve the refractive outcome theoretically.14 However, in this previous study conventional eye models were used for IOL power calculation and only the intra-operative measurement replaced pre-operative ACD measurements.

Aim of this study is to observe, whether the postoperative refractive outcome could be improved theoretically by using both pre- and intra-operative measurements for retrospective IOL power calculation with new eye models.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* Able to understand the patient information
* willing to follow the orders and coming to all follow-up visits
* willing to sign informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases that are likely to reduce the refractive outcome, such as pseudoexfoliation syndrome, traumatic cataract, severe corneal scars
* Previous ocular surgeries on the study eye
* Patients who are not able to cooperate, with eccentric fixation or insufficient ability to fixate (tremor, nystagmus)
* pregnant (pregnancy test will be taken preoperatively in women of reproductive age) or lactating women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited by the clinical investigators in the Hanusch Hospital. Each subject has to meet the inclusion and exclusion criteria and to sign informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
spherical equivalent in diopters between groups | 8 weeks postoperatively

SECONDARY OUTCOMES:
Anterior chamber depth changes in mm between intra-operative OCT measurements and 1h post-operative ACD measurements | 1 hour postoperatively
Influence of the lens thickness on IOL power calculation | 8 weeks postoperatively
Influence of post-operative tilt in degrees and decentration in mm on IOL power calculation | 8 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof Dr, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Austria